CLINICAL TRIAL: NCT02442011
Title: Hematology Biobank: In Vitro Study of Blood Disorders
Status: Recruiting | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: New York Blood Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-2918
Record Dates: First submitted 2015-05-07; First posted 2015-05-13 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hematological Disorders
Keywords: Hematology Biobank
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be processed fresh or frozen and stored in cryo vials at -80°C for future isolation of DNA. DNA isolation will be done using commercially available kits such as Applied Biosystems' "DNA Isolation from Fresh and Frozen Blood, Tissue Culture" http://tools.lifetechnologies.com/content/sfs/manuals/cms_041387.pdf Plasma needed for biomarkers analysis we be obtained from whole blood samples. Whole blood will be spun down, plasma and sediment will be separated and stored in cryo vials at -80°C. Red cells and platelets will be stored at 4C. Red cell hemolysate may be stored at 4C or stored in cryo vials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a biorepository of blood specimens from subjects with different Hematological disorders.

DETAILED DESCRIPTION:
There has been a marked increase in our knowledge of Blood Disorders in the last decade. Much of this knowledge comes from examining blood specimens from patients and subjecting these samples to red cell, plasma, serum or DNA analyses. The study team proposes to set up a Hematology biobank, which will include patient histories, their medical progress and a linked but de-identified bank of blood samples. This will enable researchers to have a large database, which can be used to learn more about these diseases.

The Hematology biobank will use whole blood, red blood cells, plasma, serum and/or DNA. Whole blood specimens, which by definition include the white cells that contain DNA, will be collected and stored in the biobank repository at the Institute for Clinical and Translational Research (ICTR) for future studies.

Blood samples will be obtained from two sources:

1. Leftover/discarded whole blood samples that were obtained for standard of care.
2. Blood samples consisting of 1-5 tubes (3-20 ml of whole blood) from patients with written consent. When possible, these samples will be obtained during routine blood draws performed for a typical visit. It may be necessary to ask patients to specifically donate blood for the study.

ELIGIBILITY:
Inclusion Criteria:

* Above 12 years of age and referred to the Hematology Division at Montefiore-Einstein
* Under the care of a Montefiore-Einstein hematologist for a hematologic disorder

Exclusion Criteria:

- Do not meet the Inclusion Criteria listed above

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Adult and pediatric patients 12 years of age and older
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Biobank | 5 years
  To have specimens available for IRB approved studies

CONTACTS AND LOCATIONS:
Overall Officials: Henny Billett, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No